CLINICAL TRIAL: NCT06554522
Title: Pragmatic Evaluation of Therapies to Enhance Respiratory Management in Preterm Infants in Africa
Brief Title: Pragmatic Evaluation of Respiratory Distress Syndrome Treatment in Africa
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Open Philanthropy (Other)
Responsible Party: Principal Investigator, Osayame Ekhaguere, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22326
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; RDS of Prematurity; Surfactant Deficiency Syndrome Neonatal; Premature Birth
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Pulmonary Atelectasis; Premature Birth | interventions — Surface-Active Agents

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-LISA Group (No Intervention): Preterm infants with respiratory distress syndrome who are on continuous positive airway pressure support and being treated with caffeine citrate.
- LISA Group (Experimental): Preterm infants with respiratory distress syndrome, who are on continuous positive airway pressure support are treated with caffeine citrate and surfactant through the less invasive surfactant administration technique.
  Interventions: Drug: Surfactant

INTERVENTIONS:
Drug: Surfactant — Surfactant is instilled into the lungs through a thin catheter passed into the trachea during laryngoscopy while on continuous positive airway pressure (CPAP)
  Other Names: Less Invasive Surfactant Administration Technique
  Arms: LISA Group

SUMMARY:
The goal of this pragmatic clinical trial is to learn if the drug surfactant given by a less invasive technique works to treat respiratory distress in preterm infants in low- and middle-income African countries where invasive ventilators are unavailable. It will also learn about the safety of the less invasive surfactant administration (LISA) technique. The main questions it aims to answer are:

Does surfactant given by a less invasive surfactant administration technique improve survival in preterm infants in low- and middle-income countries? What medical problems do participants have when receiving surfactant given by the less invasive surfactant administration technique?

Researchers will implement the less invasive surfactant administration technique and see if it works to treat respiratory distress in preterm infants compared to preterm who did not receive surfactant.

Participants with respiratory distress who are being treated with continuous positive airway pressure and caffeine citrate will:

Receive surfactant replacement therapy by the less invasive surfactant administration technique.

Be monitored for complications Be followed throughout their hospitalization to determine their survival rate.

DETAILED DESCRIPTION:
The low- and middle-income countries of Sub-Saharan Africa (SSA) carry the highest burden of preterm births and deaths. A primary driver of preterm mortality in SSA is respiratory distress syndrome. Surfactant replacement therapy by the less invasive surfactant administration (LISA) is a technique where the surfactant is administered to a preterm neonate with respiratory distress syndrome managed on continuous positive airway pressure (CPAP), reducing the need for using an invasive mechanical ventilator. In high-income countries, LISA has been shown to be effective in reducing the need for invasive mechanical ventilators and mortality. However, the impact of LISA is unknown in low-resourced settings without ventilators.

The central hypothesis is that implementing LISA in newborn units that care for preterm neonates using standardized CPAP and caffeine citrate will improve survival in preterm neonates.

PICO Outline:

Population: Preterm neonates 750 and 2000 grams or gestational age between 24- and 35 weeks at birth with respiratory distress defined by a Silverman Anderson Score of ≥5, who are spontaneously breathing and on CPAP.

Intervention: Surfactant administered through the less invasive surfactant administration (LISA), technique.

Comparator: Standard of care - standardized CPAP and Caffeine.

Outcome measures: Primary Outcome: All-cause in-hospital survival.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight between 750 and 2000 grams or gestational age between 24- and 35 weeks.
* Silverman Anderson Score ≥5 before or after CPAP treatment.
* Admitted to a study site within 24 hours of life.

Exclusion Criteria:

* Major congenital or genetic anomalies.
* Active pulmonary hemorrhage.
* Major craniofacial anomalies that preclude the successful use of CPAP

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1512 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Survival | Through hospitalization, an average of 6 months
  Survival to hospital discharge

SECONDARY OUTCOMES:
Incidence of major preterm neonatal morbidity | Through hospitalization, an average of 6 months
  Intraventricular hemorrhage, Retinopathy of Prematurity, Bronchopulmonary Dysplasia, Surgical Necrotizing Enterocolitis and Culture Positive Sepsis
The incidence of pneumothorax | Through hospitalization, an average of 6 months
  Air leaks into the space between your lung and chest wall
Hospital survival at seven day | 7 days following birth
  Survival rates assessed at day seven of life

CONTACTS AND LOCATIONS:
Overall Officials: Osayame A Ekhaguere, MBBS, MPH, Principal Investigator — Indiana University; Helen Nabwera, BMedSci, Principal Investigator — Aga Khan University; Olufunke Bolaji, MBBS, Principal Investigator — Afe Babalola University; Edgardo Szyld, MD, MS, Principal Investigator — Indiana University
Locations (8):
- Centre Hospitalier Universitaire Communautaire, Bangui, Central African Republic
- Ghana (3):
  - Korle-Bu Teaching Hospital, Accra
  - Komfo Anokye Teaching Hospital, Kumasi
  - Tamale Teaching Hospital, Tamale
- Kenya (2):
  - Coast General Teaching & Referral Hospital, Mombasa
  - Mama Lucy Kibaki Hospital, Nairobi
- Nigeria (2):
  - Federal Teaching Hospital Ido-Ekiti, Ido-Ekiti, Ekiti State
  - University of Ilorin Teaching Hospital, Ilorin, Kwara State

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest. The data shared will be coded, with no personal health information included. Approval of the request and execution of all applicable agreements (e.g., a material transfer agreement) are prerequisites to sharing data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact ***